CLINICAL TRIAL: NCT03737045
Title: Developing a Patient-centered Patient Decision Aid for Psoriasis and/or Psoriatic Arthritis Using Design Thinking.
Brief Title: Psoriatic Arthritis and Psoriasis Treatment Decision Aid
Acronym: DA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 831515
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis; Psoriasis
Keywords: Decision Aid; Shared Decision-Making
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Patients and providers will use a web-based or paper decision aid. They will not be assigned to specific arms or undergo randomized treatment.
Masking Description: Participants will have a choice of decision aids (web or paper) and will not be blinded. The study team will be aware of each prototype and decision aid that participants use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid Testing (Other): Participants will have the opportunity to test the different decision aid prototypes while selecting new treatment/therapy.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Participants will test decision aid prototypes that are designed to assist them in choosing a medication.

SUMMARY:
The purpose of this study is to create and test a patient decision aid that facilitates the shared decision-making process when patients with psoriasis and/or psoriatic arthritis are starting or switching to a new therapy.

DETAILED DESCRIPTION:
Prior to the interventional study, we will develop a decision aid using design thinking. In this interventional study, we will implement and test a patient-centered decision aid for therapy selection among patients with psoriasis and/or psoriatic arthritis who are starting or switching to a new medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of psoriasis (as confirmed by dermatologist) or psoriatic arthritis (as confirmed by rheumatologist)
3. Treated at Penn

   In addition to the above, for the observation and implementation phases of the study:
4. Initiation of a new psoriasis or psoriatic arthritis treatment

   * Biosimilars that have been approved by the FDA and available on the US market will similarly be eligible for participation
   * Patients may be taking other traditional DMARDs.
   * A washout period is not required.

Exclusion Criteria:

1. Unable to give informed consent
2. Youth, under the age of 18 years
3. Patients without psoriasis or psoriatic arthritis
4. Not being treated at a Penn clinic

   In addition to the above, for the observation and implementation phases of the study:
5. Not starting or switching to a new medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient and provider self-reported perceptions of the decision aid as measured by satisfaction survey | Up to 24 months
  Satisfaction survey to rate the decision aid and shared decision-making process

SECONDARY OUTCOMES:
Number of times decision aid was used in consultation for patients switching therapies or starting a new treatment. | Up to 24 months
  Rates of of the decision aid use

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be used to create the decision aids which will then be made available to patients, researchers, and medical centers. Physicians and researchers may request de-identified data from the PI and research plans will be reviewed on a case by case basis.